CLINICAL TRIAL: NCT06418074
Title: Effects of Exogenous Ketosis on Renal Function, Renal Perfusion, and Sodium Excretory Capacity in Patients With Essential Hypertension
Brief Title: Effects of Exogenous Ketosis on Renal Function, Renal Perfusion, and Sodium Excretory Capacity
Acronym: (KETO-HT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TZL-1-2024
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Ketosis; Essential Hypertension
Keywords: Natriuresis; Kidney circulation; Kidney physiology; Glomerular Filtration Rate
MeSH Terms: conditions — Ketosis; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone Monoester (KE4), then Placebo drink (Active Comparator): For five days each subject will receive beta-hydroxybutyrate boned to R 1,3 Butandiol (KE4), then crossed over to receive placebo drink for 5 days.
  Interventions: Dietary Supplement: Ketone Monoester (KE4); Other: Placebo
- Placebo drink, then Ketone Monoester (KE4) (Placebo Comparator): For five days each subject will receive a placebo drink three times daily, then subjects are crossed over to receive beta-hydroxybutyrate boned to R 1,3 Butandiol (KE4).
  Interventions: Dietary Supplement: Ketone Monoester (KE4); Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Monoester (KE4) — Each subject will receive beta-hydroxybutyrate boned to R 1,3 Butandiol (KE4) 300mg/kg x 3 for five days. After the treatment period effect variables will be examined.
Other: Placebo — Each subject will receive a placebo drink 3 x day for five days. After the treatment period effect variables will be examined.

SUMMARY:
This is a randomized, placebo-controlled, double-blinded crossover design. Nineteen patients with essential hypertension will be randomized to receive either ketone bodies (KE4) or placebo delivered by KetoneAid. After a period of 5-days treatment, effect variables will be measured (experiment day 1). After a washout period of 14 days, the subjects are crossed over to a similar treatment period with the other treatment. The study is terminated by measuring effect variables after the second treatment period (experiment day 2).

DETAILED DESCRIPTION:
Background: Renewed interest in ketone bodies has emerged, partly driven by the recent success of selective sodium glucose co transporter 2 (SGLT-2) inhibition in preventing cardiovascular deaths in patients with diabetes mellitus (DM) and chronic kidney disease (CKD). Effects of ketosis are of importance in order to understand the beneficial effects of SGLT-2 inhibitors and to account for the full therapeutic potential of this treatment.

Hypothesis: Ketosis decreases 24 hour systolic blood pressure and increases renal blood flow and glomerular filtration rate (GFR).

Methods: It is a randomized, placebo-controlled double-blinded cross over study. Nineteen patients with essential hypertension will be randomized to receive either ketone bodies (KE4) or for 5 days. After a wash out period of at least 14 days, the subjects are crossed over to receive the other treatment. After each treatment period effect variables will be measured including Technetium(Tc)99m - Diethylenetriamine pentaacetate (DTPA) clearance and water based positron emission tomography computed tomography (PET/CT)

Perspectives: The study has the potential to provide information regarding the therapeutic potential of treatment with ketone bodies and understanding of conditions characterized by ketosis, such as SGLT2-inhibitor treatment.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension (treatment with maximum 2 antihypertensive drugs)
* eGFR > 60ml/min
* BMI < 35 kg/m2
* Urine Albumin Creatinin Ratio (UACR) < 300mg/g
* Safe contraception if women in childbearing age

Exclusion Criteria:

* Diabetes type 1 or 2
* Heart Failure
* Pregnancy or breast feeding
* Liver disease
* Malignant disease
* Recent acute myocardial infarction (AMI), apoplexia/transient ischemic attack (TIA) (within 12 months of inclusion)
* Daily use of prescription drugs (expect for contraceptives)
* Alcohol or drug abuse
* Periodic fasting
* Routinely intake of ketogenic diet
* Treatment with immunosuppressants or SGLT2-inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-09-11 (Actual); Primary Completion 2025-06-19 (Actual); Study Completion 2025-06-19 (Actual)

PRIMARY OUTCOMES:
24-hour systolic blood pressure | Measured after each treatment period (each treatment period is 6 days)
  Change in systolic 24-hour blood pressure

SECONDARY OUTCOMES:
Renal Blood Flow (RBF) | Measured after each treatment period (each treatment period is 6 days)
  Change in RBF determined by water based PET/CT scans
GFR | Measured after each treatment period (each treatment period is 6 days)
  Change in GFR measured by Tc99m-DTPA clearance
Vasoactive hormones | Measured after each treatment period (each treatment period is 6 days)
  Change in plasma levels of aldosterone, renin, brain natriuretic peptide (BNP), atrial natriuretic peptide (ANP), copeptin
P-Beta-hydroxybutyrate | Measured after each treatment period (each treatment period is 6 days)
  Change ind p-beta-hydroxybutyrate concentration
Plasma concentration of renal tubular transport proteins | Measured after each treatment period (each treatment period is 6 days)
  Urine excretions of aquaporin 2 (AQP2), thiazide-sensitive sodium-chloride cotransporter (NCC) and distal epithelial sodium channel (ENaC)

CONTACTS AND LOCATIONS:
Overall Officials: Trine Z Lyksholm, MD, Principal Investigator — The University Clinic for Nephrology and Hypertenion, Regional Hospital Godstrup
Locations (1):
- The University Clinic in Nephrology and Hypertension, Gødstrup Region Hospital, Herning, Denmark

IPD SHARING:
Plan to Share IPD: No